CLINICAL TRIAL: NCT00145041
Title: An Evaluation of the Pharmacokinetic Profile of VSLI (Vincristine Sulfate Liposome Injection, 0.16 mg/mL) in Patients With Malignant Melanoma and Hepatic Dysfunction Secondary to Metastases
Brief Title: Pharmacokinetic Study of Liposomal Vincristine in Patients With Malignant Melanoma & Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VSLI-12-HEPHARM
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2012-01-05 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VSLI (Experimental): Single armed study; all subjects received VSLI
  Interventions: Drug: Vincristine Sulfate Liposomes Injection

INTERVENTIONS:
Drug: Vincristine Sulfate Liposomes Injection — Marqibo (VSLI) 1.0 mg/m2 delivered by intravenous infusion over 1 hour every 2 weeks.
  Other Names: Marqibo

SUMMARY:
The purpose of this study is to see how vincristine, when placed in an oil droplet called a liposome (VSLI), is absorbed, distributed (moved around) and excreted from the the body (pharmacokinetics). This study will also assess the safety of VSLI and to see if VSLI will slow the growth or shrink tumors in patients with metastatic melanoma that has resulted in liver impairment, and who have relapsed after previous therapies.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: To assess the pharmacokinetics of VSLI administered intravenously to patients with malignant melanoma and hepatic dysfunction secondary to metastases.

Secondary: To assess the safety and antitumor activity of VSLI in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, surgically nonresectable Stage III or IV metastatic cutaneous, mucosal, or choroidal melanoma, and not be eligible for a treatment protocol of a higher priority.
* Patients must have secondary tumor involvement of the liver confirmed by CT scan and a bilirubin level of 1.6-3.0 mg/dL (National Cancer Institute, Common Terminology Criteria for Adverse Events Grade 2) (MD Anderson Cancer Center normal range is 0-1.0 mg/dL).
* Patients must have bidimensionally measurable disease.
* Patients with nonchoroidal melanoma must have received prior chemotherapy for metastatic disease with cytotoxic or biological drugs. Patients with choroidal melanoma may or may not have received prior chemotherapy for metastatic disease with cytotoxic or biological drugs.
* Patients must have a Performance Status of 0, 1, 2, or 3 (Zubrod Scale).
* Patients must have recovered from the adverse effects of prior chemotherapy (including cytotoxic agents and biological response modifiers), and/or irradiation therapy.
* Patients must have an absolute neutrophil count ≥1.0 x 10*9/L and a platelet count of ≥100 x 10*9/L.
* Patients must have adequate renal function demonstrated by a creatinine level of ≤2.0 mg/dL.
* Patients must have a life expectancy of >8 weeks.
* Patients must provide a signed informed consent document indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.

Exclusion Criteria:

* Patients treated with radiotherapy, chemotherapy, immunotherapy, vaccine treatment and/or alternative anticancer treatments (including investigational drugs) within 3 weeks prior to study enrollment.
* Patients treated with hepatic chemo-embolization within 4 weeks prior to study enrollment.
* Patients with severe hepatic impairment demonstrated by plasma ammonia levels >105 mMol/L or serum albumin <2.0 g/dL or serum bilirubin >3.0 mg/dL.
* Patients with serious intercurrent illness.
* Patients who have had major surgery within 4 weeks of enrollment.
* Patients with advanced symptomatic central nervous system (CNS) involvement by melanoma and those on phenytoin or requiring steroids for brain metastases, spinal cord compression, or meningeal "carcinomatosis".Patients with asymptomatic and stable metastatic CNS disease can be enrolled.
* Patients receiving treatment with phenytoin and/or corticosteroids within 1 week of enrollment. Patients must remain off of these medications for the duration of the treatment phase of the study.
* Patients with a history of neurological disorders unrelated to chemotherapy (including familial neurological diseases and acquired demyelinating disorders).
* Patients with Grade 3 or greater sensory, motor or autonomic neuropathy at screening from any cause.
* Patients receiving treatment with drugs known to inhibit or induce hepatic drug metabolism by cytochrome P450-3A4 isoenzymes and/or P-glycoprotein within 1 week of study enrollment. Patients must remain off of these drugs until the collection of the Cycle 4 pretreatment PK sample.
* Patients with past or current history of liver parenchymal or hepatobiliary disease unrelated to cancer (including but not limited to conditions such as liver cirrhosis, acute/chronic hepatitis, ascending cholangitis, etc).
* Patients who are pregnant or lactating. Females of childbearing potential must have a negative urine or blood pregnancy test at screening. Both men and women must be practicing an adequate method of birth control for the duration of the study. Acceptable methods of birth control include use of an intrauterine device (IUD), oral contraceptive pills, implanted, transdermal, or injected contraceptives, barrier methods with spermicide, and abstinence.
* Patients who are unable to return for follow up re-evaluation and assessment of response to VSLI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-02; Primary Completion 2007-09 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agop Bedikian, MD, Principal Investigator — MD Anderson Cancer Center, Dept of Melanoma
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center, open-label, single-arm, Phase 1 study to assess the PK of VSLI in subjects with malignant melanoma and hepatic dysfunction secondary to liver metastases.
Pre-assignment Details: Eligible subjects were to have liver metastases confirmed by computed tomography (CT) scan at screening. Categorization of hepatic dysfunction at screening included Child-Pugh System.
Groups:
- Overall Study: This was a non-randomized, open-label, single arm, single-center Phase 1 study. All subjects received the same treatment. All subjects received Marqibo (VSLI) 1.0 mg/m2 delivered by intravenous infusion over 1 hour every 2 weeks.
Period: Overall Study
Arm/Group | Overall Study
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: T 1/2
Description: The PK profiles of total plasma VCR following a single intravenous infusion at a target dose of 1.0 mg/m2 for approximately 1 hour every 2 weeks (one cycle) to three male and four female subjects with malignant melanoma and hepatic dysfunction secondary to metastases were measured.
Time Frame: cycle 1 day 1
Population: all patients enrolled
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Overall Study
Number analyzed (Participants) | 7
hr | 9.94 (1.22)

2. Primary Outcome: Clearance
Description: The pharmacokinetic profile of VCR on Day 1 of Cycle 1 Cl is mL/h/m2
Time Frame: Day 1 of Cycle 1
Population: All subjects enrolled
Measure: Mean (Standard Deviation); unit: ml/h/m2
Arm/Group | Overall Study
Number analyzed (Participants) | 7
ml/h/m2 | 193 (80.3)

3. Primary Outcome: Volume of Distribution
Description: The PK profiles of total plasma VCR following a single intravenous infusion at a target dose of 1.0 mg/m2 for approximately 1 hour
Time Frame: cycle 1 day 1
Population: all patients enrolled
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Overall Study
Number analyzed (Participants) | 7
mL/m2 | 2722 (1066)

ADVERSE EVENTS:
Time Frame: The AE reporting period for this study was from the time of the first dose of VSLI until 30 days after the last dose of VSLI.
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 7/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=7)
Cardiac arrest (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Malignant melanoma (Skin and subcutaneous tissue disorders) | 3 (3) — Disease progression of melanoma
Ascites (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (General disorders) | 1 (1) — Pain, right upper quadrant
Disease progression (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study (N=7)
Malignant melanoma (Skin and subcutaneous tissue disorders) | 4 (4)
Fatigue (General disorders) | 4 (4)
Decreased appetite (General disorders) | 4 (4)
Ascites (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (General disorders) | 3 (3)
Oedema, peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)
Anxiety (Nervous system disorders) | 2 (2)
Insomnia (General disorders) | 2 (2)
Abdominal distention (General disorders) | 1 (1)
Abdominal pain, upper (General disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Gait disturbance (Nervous system disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Hypomagnesaemia (General disorders) | 1 (1)
Hyponatraemia (General disorders) | 1 (1)
tumor pain (General disorders) | 1 (1)
confusional state (Nervous system disorders) | 1 (1)
depression (Nervous system disorders) | 1 (1)
sleep disorder (General disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
anaemia (Blood and lymphatic system disorders) | 1 (1)
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
drug hypersensitivity (General disorders) | 1 (1)
seasonal allergy (General disorders) | 1 (1)
blood bilirubin increased (Hepatobiliary disorders) | 1 (1)
weight increased (General disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1)
hyperbilirubinaenemia (Hepatobiliary disorders) | 1 (1)
central line infection (Infections and infestations) | 1 (1)
neuropathy, peripheral (Nervous system disorders) | 1 (1)
night sweats (General disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
menopause (General disorders) | 1 (1)
hypotension (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The dose administered to subjects with impaired liver function was ~1 mg/m2 which is lower than is administered to subjects with normal liver function (2 mg/m2). The impact of liver impairment on that higher dose remains unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less